CLINICAL TRIAL: NCT03270020
Title: Evaluation of Efficacy of Denosumab in Adult Patients With Langerhans Cell Histiocytosis (LCH): a Multiple-site, Single Arm, Open Label Clinical Trial
Brief Title: Denosumab for the Treatment of Adult LCH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hellenic Society for the Study of Bone Metabolism (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20159460
Record Dates: First submitted 2017-08-26; First posted 2017-09-01 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Langerhans Cell Histiocytosis
Keywords: treatment; denosumab; Positron Emission Tomography (PET) CT scan
MeSH Terms: conditions — Histiocytosis, Langerhans-Cell | interventions — Denosumab

STUDY DESIGN:
Intervention Model Description: The investigational arm will recruit patients who will receive denosumab 120mg sc every 2 months. The estimated duration of the recruitment period is 12 months.
  The treatment period would be 6 months (denosumab administration on months: 0, 2, 4, 6) and the follow-up period would be 12 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): This is a single arm study; the study arm include all patients participating in the study who will all receive Denosumab 70 MG/ML [Xgeva]
  Interventions: Drug: Denosumab 70 MG/ML [Xgeva]

INTERVENTIONS:
Drug: Denosumab 70 MG/ML [Xgeva] — As already described in arm description
  Other Names: Xgeva

SUMMARY:
This study is aiming to evaluate the efficacy of denosumab among adult patients suffering from Langerhans Cell Histiocytosis (LCH).

DETAILED DESCRIPTION:
The majority and diversity of clinical manifestations in LCH are attributed to immunological dysfunction resulting from langerhans cell (LC) derived cytokine secretion both at the lesional and systemic level. In a recent study, Receptor Activator of Nuclear Factor Kappa-B Ligand (RANKL) was found to be abundantly expressed in cells within diverse LCH lesions from adult patients, especially in inflammatory infiltrates, a finding in line with a previously reported high osteoprotegerin (OPG) and low RANKL levels in the serum of patients with or without bone involvement. RANKL expression was associated with concomitant p65 Nuclear Factor Kappa-B (NFκB) nuclear staining, the main downstream effector of RANKL signaling, suggesting that lesional cell activation may be triggered locally by RANKL. Combining the serum and the lesional results, it can be inferred that there is an ongoing process of countervailing OPG production against lesional RANKL, which could be one of the self defense mechanisms among LCH patients. Therefore, the use of denosumab seems a rational treatment option in LCH in order to support and enhance the defensive OPG action and hopefully control or even interrupt the lesional immunological process.

The primary study objective is to assess the therapeutic efficacy of denosumab 120 mg every 8 weeks (Q8W) sc in adult LCH patients.

Secondary Objectives:

1. To define an uniform treatment approach for LCH patients with mild symptoms and low risk disease.
2. To explore the efficacy of denosumab 120 mg Q8W sc in reducing disease reactivations after treatment completion.
3. To illustrate the safety profile of denosumab in LCH patients. The primary efficacy endpoint is defined as the percentage of patients with progression of disease at Month 8.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18 years of age)
* Definitive diagnosis of LCH [Based on clinic-pathological evidence with microscopic examination and at least one of the following immunological staining: Langerin (CD 207) positivity, Cluster of Differentiation 1a (CD1a) positivity, Presence of Birbeck granules on electronic microscopy]
* Mild symptoms (symptoms of low intensity; no need for hospitalization) and low risk disease needing first line systemic therapy for LCH because of:

  * single system disease with multifocal lesions, or
  * single system disease with "special site" lesions (vertebral lesions with intraspinal extension, craniofacial bone lesions with soft tissue extension), or
  * multi-system disease without involvement of risk organs [hematopoietic system, spleen, liver, tumorous central nervous system (CNS)].
* Have signed the informed consent form (consent should be taken before any study-specific procedure is performed).
* A patient should undergo a PET-CT imaging test, in order for him to be deemed suitable for the study. The initial PET-CT either may have been carried out, within 3 months prior to visit 1, regardless of the diagnostic center or the type of the device, which has been used for, or may take place in the context of visit 2, at the diagnostic center(s) specialized on Nuclear Medicine, which have been partnered with the Sponsor. Whichever is the case, the initial PET-CT report should be legible and accurate, so that to be assessed by the qualified physician, responsible for the PET-CT test at the partnered diagnostic center(s).

Exclusion Criteria:

* Symptomatic multi system LCH - no risk organs involved.
* Multi-system LCH (with or without symptoms) - risk organs involved.
* Isolated pulmonary LCH disease
* Previous administration of denosumab from clinical trials or other use (e.g. commercial use).
* Current participation in another clinical trial or having received any investigational product within the last 3 months.
* Impaired renal function as determined by an estimated glomerular filtration rate (eGFR) of ≤ 30 mL/min/1,73m2 [using the Chronic Kidney Disease-Epidemiology, (CKD-EPI) formula].
* Patients that have received oral bisphosphonates within 6 months of study enrollment or intravenous bisphosphonates, fluoride and strontium ranelate within 1 year of study enrollment.
* Treatment with immune suppressive agents within 4 weeks from baseline evaluation.
* Patients with severe impairment of clinical condition including: severely impaired pulmonary function [for example total lung capacity (TLC)<60%, forced expiratory volume 1 (FEV1)<30%, diffusing capacity of the lungs for carbon monoxide (DLCO)<30%, partial pressure of oxygen (PaO2)<55 mmHg), long term oxygen therapy or cor pulmonale.
* Known to have a liver failure or chronic hepatic disease e.g. cirrhosis, chronic hepatitis; or elevated transaminases defined as alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) > 2 fold the upper limit of normal laboratory range.
* Heart failure [New York Heart Association (NYHA) Functional Classification above 2].
* Patients with life expectancy of less than one year.
* Female subjects of childbearing potential who refuse to use a reliable contraceptive method throughout the study, defined as use of 2 highly effective forms of contraception and continuation of use for 7 months after last administration of study drug. Birth control methods that can achieve a failure rate of less than 1% per year, when used consistently and correctly, are considered as highly effective.
* Pregnancy, planning a pregnancy or currently lactating
* Severe concurrent illness which in the investigator's opinion may confound patient evaluation, e.g. malignancy (except basal cell carcinoma, cervical or breast ductal carcinoma in situ) within the last 5 years.
* Known alcohol or drug abuse.
* Parathyroid hormone (PTH), PTH derivatives, teriparatide, odanacatib, anabolic steroids, testosterone, glucocorticosteroids (> 5 mg/day of prednisone equivalent for > 10 days), systemic hormone-replacement therapy, selective estrogen receptor modulators (SERMs), raloxifene, tibolone, calcitonin use within the last 6 weeks.
* Evidence of hyper- or hypothyroidism; patients with an abnormal thyroid stimulate hormone (TSH) level on thyroid treatment (patients on stable thyroid treatment with a normal TSH allowed); current hyper- or hypoparathyroidism; current hyper or hypocalcemia (hypercalcemia based on albumin adjusted serum calcium > 10.40 mg/dL; hypocalcemia based on albumin adjusted serum calcium < 8.5 mg/dL); vitamin D deficiency (25-hydroxy vitamin D level < 20 ng/mL; if the resulted value of the retest is 20 ≥ ng/Ml, after repletion with 50,000 - 100,000 IU of cholecalciferol, subject will be allowed. The retest should be carried out within 30 days post to visit 1(screening)); rheumatoid arthritis; Paget's disease; any known bone disease with osteolytic and/or osteoblastic lesions that would interfere with interpretation of findings.
* Known sensitivity to mammalian cells, denosumab or any components of denosumab 120mg, or any of the products to be administered during the study (e.g., calcium or vitamin D).
* History of any Solid Organ or Bone Marrow Transplant.
* History of osteonecrosis of the jaw, and/or recent tooth extraction or other dental surgery; or planned invasive dental work during the study.
* Intolerance to calcium supplements.
* Malabsorption syndrome; severe malabsorption including Celiac disease, Short Bowel Syndrome, Crohn's disease, Previous Gastric Bypass.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-09-07 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2025-01-14 (Actual)

PRIMARY OUTCOMES:
Primary efficacy endpoint: effect of denosumab treatment on the activity status of the disease (Incidence of patients with active disease) | 8 months
  The primary efficacy endpoint will be measured through the incidence of patients with active disease at Month 8. Given that all patients have active disease at baseline the incidence of patients with active disease at Month 8 will provide the efficacy of denosumab in controlling the disease within this time frame.

SECONDARY OUTCOMES:
Secondary efficacy endpoint: development of disease-related permanent sequelae during the study period (Incidence of disease-related permanent sequelae) | 18 months
  Incidence of disease-related permanent sequelae, developed during the study, at month 18. In specific, permanent sequelae such as diabetes insipidus, anterior pituitary deficiencies, and pulmonary failure will be assessed at the end of the study in order to evaluate the efficacy of denosumab in preventing those conditions.

OTHER OUTCOMES:
Safety endpoints: Incidence of all Adverse Events during the trial | 18 months
  Incidence of Adverse Events during the trial. In specific, all adverse events will be assessed at the end of the study period in order to evaluate the safety issues of denosumab treatment in LCH.
Safety endpoint: Incidence of all adverse events on bone metabolism following Denosumab treatment and its withdrawal | 30 months
  Assess the effects of treatment and its withdrawal on bone metabolism, in particular the presence or not of rebound of bone turnover following discontinuation of Denosumab

CONTACTS AND LOCATIONS:
Overall Officials: Polyzois Makras, MD, PhD, Principal Investigator — Dpt of Endocrinology & Diabetes, 251 Hellenic AirForce & VA General Hospital, Athens, Greece
Locations (1):
- 251 Hellenic AirForce & VA General Hospital, Dpt of Endocrinology, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Makras P, Tsoli M, Anastasilakis AD, Thanou M, Kaltsas G. Denosumab for the treatment of adult multisystem Langerhans cell histiocytosis. Metabolism. 2017 Apr;69:107-111. doi: 10.1016/j.metabol.2017.01.004. Epub 2017 Jan 12. PMID 28285639
- [Background] Makras P, Salagianni M, Revelos K, Anastasilakis AD, Schini M, Tsoli M, Kaltsas G, Andreakos E. Rationale for the application of RANKL inhibition in the treatment of Langerhans cell histiocytosis. J Clin Endocrinol Metab. 2015 Feb;100(2):E282-6. doi: 10.1210/jc.2014-2654. Epub 2014 Nov 6. PMID 25375981
- [Background] Makras P, Polyzos SA, Anastasilakis AD, Terpos E, Kanakis G, Schini M, Papatheodorou A, Kaltsas GA. Serum osteoprotegerin, RANKL, and Dkk-1 levels in adults with Langerhans cell histiocytosis. J Clin Endocrinol Metab. 2012 Apr;97(4):E618-21. doi: 10.1210/jc.2011-2962. Epub 2012 Jan 25. PMID 22278426
- [Background] Girschikofsky M, Arico M, Castillo D, Chu A, Doberauer C, Fichter J, Haroche J, Kaltsas GA, Makras P, Marzano AV, de Menthon M, Micke O, Passoni E, Seegenschmiedt HM, Tazi A, McClain KL. Management of adult patients with Langerhans cell histiocytosis: recommendations from an expert panel on behalf of Euro-Histio-Net. Orphanet J Rare Dis. 2013 May 14;8:72. doi: 10.1186/1750-1172-8-72. PMID 23672541